CLINICAL TRIAL: NCT00521066
Title: A Prospective, Multi-centre Study to Evaluate the Clinical Performance of the GYNECARE PROSIMA* Pelvic Floor Repair System as a Procedure for Pelvic Organ Prolapse
Brief Title: GYNECARE PROSIMA* Pelvic Floor Repair System for Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 300-06-005
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Prosima Pelvic Floor Repair System
  Interventions: Device: GYNECARE PROSIMA* Pelvic Floor Repair System

INTERVENTIONS:
Device: GYNECARE PROSIMA* Pelvic Floor Repair System — procedure for pelvic organ prolapse
  Other Names: mesh pelvic floor repari

SUMMARY:
The purpose of this study is to is to evaluate the success of the GYNECARE PROSIMA* system in women with symptoms for pelvic organ prolapse (POP) requiring surgical correction of POP.

(*TRADEMARK)

DETAILED DESCRIPTION:
The GYNECARE PROSIMA* system provides a simplified mesh repair, avoiding the need for dissection outside the pelvic cavity.

ELIGIBILITY:
Inclusion Criteria:

* Candidates with symptomatic pelvic organ prolapse of ICS POP-Q Stage II or III, suitable for surgical repair. Vaginal hysterectomy, perineal repair and/or mid urethral sling procedures for incontinence may be performed concurrently.
* Age ≥ 18 years.
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires, and documents this agreement by signing the Ethics Committee / IRB approved informed consent.

Exclusion Criteria:

* Additional surgical intervention concurrent to the PROSIMA procedure (e.g. sacrocolpopexy, paravaginal repair, tubal sterilisation).
* Previous repair of pelvic organ prolapse involving insertion of mesh.
* Previous hysterectomy within 6 months of scheduled surgery.
* Experimental drug or experimental medical device within 3 months prior to the planned procedure.
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Coagulation disorder or on therapeutic anticoagulant therapy at the time of surgery.
* History of chemotherapy or pelvic radiation therapy.
* Systemic disease known to affect bladder or bowel function (e.g. Parkinson's disease, multiple sclerosis, spina bifida, spinal cord injury or trauma).
* Current evaluation or treatment for chronic pelvic pain (e.g. interstitial cystitis, endometriosis, coccydynia, vulvodynia).
* Nursing or pregnant or intends future pregnancy.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 with symptomatic pelvic organ prolapse of ICS POP-Q Stage II or III, suitable for surgical repair
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Success based on overall POP-Q score at 12 months post-procedure. | 12-months
  Success is determined by achievement of an overall POP-Q score of ICS Stage ≤1, without further re-intervention for POP.

SECONDARY OUTCOMES:
Success based on overall POP-Q score at 24 months post-procedure. | 24 months
  Success is determined by achievement of an overall POP-Q score of ICS Stage ≤1, without further re-intervention for POP
Success based on treated compartment ICS POP-Q stage | 12 months
  Success will be determined by achievement of treated compartment POP-Q score of ICS Stage ≤1, without further re-intervention for POP.
Success based on treated compartment ICS POP-Q stage | 24 months
  Success will be determined by achievement of treated compartment POP-Q score of ICS Stage ≤1, without further re-intervention for POP.
Success defined as the leading edge within the hymen | 12 months
  Success defined as the leading edge within the hymen (i.e. all POP-Q values to be less than 0, without further re-intervention for POP)
Success defined as the leading edge within the hymen | 24 months
  Success defined as the leading edge within the hymen (i.e. all POP-Q values to be less than 0, without further re-intervention for POP)
Mean PFDI-20 score | 12 months
Mean PFDI-20 score | 24 months
Mean change from baseline in PFDI-20 scores | 24 months
Mean change from baseline in PFDI-20 scores | 12 months
Mean POPDI score | 12 months
  POPDI is a sub score of PFDI-20
Mean POPDI score | 24 months
  POPDI is a sub score of PFDI-20
Mean change from baseline in POPDI score | 12 months
  POPDI is a sub scores of PFDI-20
Mean change from baseline in POPDI score | 24 months
  POPDI is a sub score of PFDI-20
Mean CRADI score | 12 months
  CRADI is a sub score of PFDI-20
Mean CRADI score | 24 months
  CRADI is a sub score of PFDI-20
Mean change from baseline in CRADI score | 12 months
  CRADI is a sub score of PFDI-20
Mean change from baseline in CRADI score | 24 months
  CRADI is a sub score of PFDI-20
Mean UDI score | 12 months
  UDI is a sub score of PFDI-20
Mean UDI score | 24 months
  UDI is a sub score of PFDI-20
Mean change from baseline in UDI score | 12 months
  UDI is a sub score of PFDI-20
Mean change from baseline in UDI score | 24 months
  UDI is a sub score of PFDI-20
EuroQol (EQ-5D health state) change from baseline | 12 months
EuroQol (EQ-5D health state) change from baseline | 24 months
Mean PFIQ-7 score | 12 months
Mean PFIQ-7 score | 24 months
Mean change from baseline in PFIQ-7 score | 12 months
Mean change from baseline in PFIQ-7 score | 24 months
Mean POPIQ score | 12 months
  POPIQ is a sub-score of PFIQ-7
Mean POPIQ score | 24 months
  POPIQ is a sub-score of PFIQ-7
Mean change from baseline in POPIQ score | 12 months
  POPIQ is a sub-score of PFIQ-7
Mean change from baseline in POPIQ score | 24 months
  POPIQ is a sub-score of PFIQ-7
Mean CRAIQ score | 12 months
  CRAIQ is a sub-score of PFIQ-7
Mean CRAIQ score | 24 months
  CRAIQ is a sub-score of PFIQ-7
Mean change from baseline in CRAIQ score | 12 months
  CRAIQ is a sub-score of PFIQ-7
Mean change from baseline in CRAIQ score | 24 months
  CRAIQ is a sub-score of PFIQ-7
Mean UIQ score | 12 months
  UIQ is a sub-score of PFIQ-7
Mean UIQ score | 24 months
  UIQ is a sub-score of PFIQ-7
Mean change from baseline in UIQ score | 12 months
  UIQ is a sub-score of PFIQ-7
Mean change from baseline in UIQ score | 24 months
  UIQ is a sub-score of PFIQ-7
Mean PISQ-12 score | 12 months
  In subjects sexually active at baseline, assessment of sexual function
Mean PISQ-12 score | 24 months
  In subjects sexually active at baseline, assessment of sexual function
Mean change from baseline in PISQ-12 score | 12 months
  In subjects sexually active at baseline, assessment of sexual function
Mean change from baseline in PISQ-12 score | 24 months
  In subjects sexually active at baseline, assessment of sexual function
Incidence of new onset dyspareunia, resolution or continuance of pre-existing dyspareunia | ongoing
Length of procedure | perioperative
  From time to first incision to time of last suture used to secure VSD
Pain score measured using Visual Analog Scale (VAS). | 24 hours post surgery and at the 3-4 week visit
Discomfort of balloon removal, measured using VAS at time of removal. | 24 hrs post-surgical
Subject perception of VSD: Awareness | 3-4 week visit
  Measured by visual analogue scale
Subject perception of VSD: Discomfort | 3-4 week visit
  Measured by visual analogue scale
Subject perception of VSD: Acceptability of discharge | 3-4 week visit
  Measured by visual analogue scale
Subject global impression | 12 month visit
  assessed on a 5 point Likert scale
Subject global impression | 24 month visit
  assessed on a 5 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, M.D., Study Director — Ethicon, Inc.
Locations (11):
- United States (5):
  - Specialists in Urology, Naples, Florida
  - Female Pelvic Medicine and Urogynecology Institute of Michigan, Dearborn, Michigan
  - Female Pelvic Medicine & Urogynecology, Grand Rapids, Michigan
  - The Institute for Female Pelvic Medicine & Reconstructive Surgery, Allentown, Pennsylvania
  - Magee Women's Hospital of the Universtiy of Pittsburgh, Pittsburgh, Pennsylvania
- Royal Women's Hospital, Melbourne, Australia
- Germany (2):
  - Bereich Urogynakologie, Halle
  - Universitatsklinik Tubingen, Tübingen
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - North Hampshire Hospital, Hampshire
  - St. Mary's Hospital, Manchester

REFERENCES:
- [Result] Zyczynski HM, Carey MP, Smith AR, Gauld JM, Robinson D, Sikirica V, Reisenauer C, Slack M; Prosima Study Investigators. One-year clinical outcomes after prolapse surgery with nonanchored mesh and vaginal support device. Am J Obstet Gynecol. 2010 Dec;203(6):587.e1-8. doi: 10.1016/j.ajog.2010.08.001. PMID 20934681
- [Result] Sayer T, Lim J, Gauld JM, Hinoul P, Jones P, Franco N, Van Drie D, Slack M; Prosima Study Investigators. Medium-term clinical outcomes following surgical repair for vaginal prolapse with tension-free mesh and vaginal support device. Int Urogynecol J. 2012 Apr;23(4):487-93. doi: 10.1007/s00192-011-1600-3. Epub 2011 Dec 6. PMID 22143448